CLINICAL TRIAL: NCT00551798
Title: Prediction of the Response to Chemotherapy by Tomoscintigraphie the MIBI in the Balance Sheet Pre Hodgkin's Disease and Lymphoma Malins High Grade
Acronym: MIBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I04016
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2005-03

CONDITIONS: Hodgkin's Disease; Malignant Lymphomas High Grade; Chemoresistance
Keywords: Hodgkin's Disease; Malignant lymphomas high grade; Chemoresistance; MIBI; PGP; MRP1; Tumor response
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: TEP au MIBI — Intravenous injection of MIBI.The review lasted 30 min, during which the patient should not move.

SUMMARY:
Predicting response to chemotherapy in patients with Hodgkin's disease or lymphoma high-grade malignant de novo or recurrence.

The non-Hodgkin's lymphoma and high-grade Hodgkin's disease may show resistance to chemotherapy, regardless of their initial extension. The failure of treatment is most often correlated with an incomplete answer or lack of response to chemotherapy as a result chemoresistance. This drug, which may involve the gene MDR1 (multidrug resistance) encoding the protein PGP, can be studied in vivo by MIBI scan. The MIBI is behind a tracer perfusionnel used routinely to explore myocardial perfusion, but it has other characteristics of fixing, which can be used in oncological imaging (fixation by glial tumors of high grade).Prospective Study, which includes conducting a tomoscintigraphie 30 minutes after injection of 20 mCi of 99mTc-MIBI in initial stock or relapse of high-grade lymphoma and Hodgkin's disease any stage (I-IV). Fixing the MIBI is compared with morphological abnormalities detected by CT and the setting of lesions by 18FDG. Patients will be treated in a traditional way, without changes in treatment protocols used in routine. Patients with a negative MIBI scan, will be watched with particular attention in order to detect insufficient response to chemotherapy. The only change, the care of patients, only for the achievement of an initial consideration of non-invasive imaging, further, which is the tomoscintigraphie the MIBI. Of the tumor samples, will be evaluated by immunohistochemistry, the expression of PGP and the MRP1 (two proteins associated with the drug). On blood, may be carried out genotyping of MDR1, MRP1 and MRP2 to the patient.

ELIGIBILITY:
Inclusion Criteria:

* initial Attainment: High-grade NHL or Hodgkin's disease all stages:I, II, III et IV.
* Relapse: High-grade NHL or Hodgkin's disease relapse in all stages:I, II, III et IV.
* Patients recruited by the Network of clinical hematology du Limousin
* Patients older than 18 years with or without brain damage

Exclusion Criteria:

* Pregnant women or nursing mothers or without effective contraception
* Patients without coverage by social security
* Patients who started steroids referred to antitumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2005-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the predictive value of fixing the MIBI by the masses lymphomatous or Hodgkiniennes (initial or repeated) on the response to chemotherapy in 4 months.

SECONDARY OUTCOMES:
• To evaluate the predictive value of fixing the MIBI on the therapeutic response at 1 month and at the end of treatment.
• To evaluate the predictive value of fixing the MIBI on disease free survival and overall survival of patients.
• To evaluate the correlation between fixing MIBI and the expression of tumor PGP and / or MDR.
• Assess the influence of tumor protein expression PGP on the MRP or disease free survival and overall patient
• Possibly, studying the influence of genotype MDR1 and MRP2 on the expression of tumor protein PGP and MRP2 and on the response to treatment at different periods.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques MONTEIL, MD, Principal Investigator — University Hospital, Limoges
Locations (5):
- France (5):
  - Anatomo-pathology, Limoges
  - Hematology, Limoges
  - Nuclear Medicine, Limoges
  - Pharmacology, Limoges
  - Radiology, Limoges